CLINICAL TRIAL: NCT01496261
Title: Comparative Pharmacokinetics of Clopidogrel 75mg and Aspirin 100mg After Single Oral Administration as a Fixed Dose Combination Versus Separate Combination in Healthy Male Volunteers
Brief Title: Comparative Pharmacokinetics Study of Clopidogrel and Aspirin Fixed-dose Combination Versus Separate Combination-2nd Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Inje University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 132HPS11I
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Coronary Artery Disease
Keywords: Clopidogrel; Aspirin; Combination; Pharmacokinetics; Phase 1
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel and Aspirin (Active Comparator)
  Interventions: Drug: Clopidogrel and Aspirin
- Coprigerl (Experimental)
  Interventions: Drug: Fixed dose combination of clopidogrel/aspirin

INTERVENTIONS:
Drug: Clopidogrel and Aspirin — Clopidogrel and Aspirin seperate combination, single dose
  Other Names: Clopidogrel: Plavix; Aspirin: Astrix
  Arms: Clopidogrel and Aspirin
Drug: Fixed dose combination of clopidogrel/aspirin — Fixed dose combination of clopidogrel/aspirin
  Other Names: Coprigrel
  Arms: Coprigerl

SUMMARY:
The purpose of this study is to compare pharmacokinetics between fixed-dose combination and separate combination of clopidogrel 75mg/aspirin 100mg.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male volunteer aged 20 to 55, and within 20% of ideal body weight.
* Have not any congenital or chronic diseases and medical symptom.
* Appropriate subject for the study judging from examinations(interview, vital signs, 12-lead ECG, physical examination, blood, urinalysis result on screening.
* Able to participate in the entire trial.
* Signed the informed consent form prior to study participation.

Exclusion Criteria:

* Take metabolic enzyme inducing or inhibiting drugs like barbiturates within 28 days prior to the first IP administration.
* show evidence of acute disease within 28 days prior to the first IP administration.
* Have the medical history of bleeding symptom or bleeding disease
* Have the disease history(ex. Inflammatory intestinal disease, stomach or duodenum ulcer, liver and bowels disease, appendectomy except of gastrointestinal surgery history) that may influence on the absorption, distribution, metabolism and excretion of the drug.
* Have relevant hypersensitivity against drug or clinically significant allergic diseases except mild rhinitis that doesn't need medication.
* Have hypersensitivity reaction histories for Clopidogrel or aspirin.
* Have abnormal laboratory result. AST or ALT > 1.25 times of upper limit/ Total bilirubin > 1.5 times of upper limit/ PT, aPTT, BT over upper limit/ Platelet count <150X10^9/L or >350X10^9/L
* A drug abuse or a heavy caffeine consumer (more than 5cups per a day) or a heavy smoker (more than 10 cigarettes per a day) or a regular alcohol consumer(more than 30g/day) or drinking within 7days prior to the first IP administration.
* Have a diet(Especially, grapefruit juice-within 7days prior to the first IP administration) that may influence on the absorption, distribution, metabolism and excretion of the drug(s).
* Have donated whole blood within 60 days prior to the first IP administration.
* Participated in the other clinical trials within 90days prior to the first IP administration.
* Take medicine which affect to this trial within 10 days prior to the first IP administration.
* Appropriate subject for the trial judging from principal investigator.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Assess the pharmacokinetic characteristics of clodiogrel/acetylsalicylic acid. | FDAAA) Pre-dose, 0.33h, 0.67h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 6h, 8h, 10h, 12h, 24h
  Assess Cmax, AUC, Tmax and t1/2(half-life) of clodiogrel/acetylsalicylic acid.

SECONDARY OUTCOMES:
Assess the pharmacokinetic characteristics of salicylic acid. | Pre-dose, 0.33h, 0.67h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 6h, 8h, 10h, 12h, 24h
  Assess Cmax, AUC, Tmax, t1/2(Half-life) of salicylic acid.

CONTACTS AND LOCATIONS:
Overall Officials: JL Ghim, Dr., Principal Investigator — Inje University
Locations (1):
- Inje University Pusan Paik Hospital, Jin-gu, Busan, South Korea